CLINICAL TRIAL: NCT04839874
Title: Health Seeking Behaviour in Women Diagnosed With Gynaecological Cancer: Can it be Modified to Improve Patient Outcomes?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: NHS Grampian
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Gynaecological Cancer
Keywords: Health seeking behaviour; Pelvic examination
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Semi-structured qualitative interviews

SUMMARY:
This study will focus on speaking to women who have been diagnosed with one of the five main gynaecological cancers: ovarian, endometrial (womb), cervical, vulval and vaginal. Too many women are dying from gynaecological cancer in the UK. There are many reasons for this, but the study investigators think that embarrassment might be one of the reasons. It can be embarrassing to talk about gynaecological cancers or the symptoms that they cause. This might lead some women to delay going to their doctor when they have symptoms. This study will speak with women who have been diagnosed with a gynaecological cancer to ask them what they did before they were diagnosed; when did they realise something was wrong; what made them go to their doctor; did having gynaecological symptoms make them think differently about going to the doctor? This information will be used to find ways of making it as easy as possible for women to go to their doctors as early as possible. This will hopefully see fewer women dying from these cancers.

DETAILED DESCRIPTION:
The study will explore the research questions using qualitative semi-structured interviews with women diagnosed with gynaecological cancer. A study information sheet, reply slip and a reply-paid envelope will be sent to eligible patients by their secondary care clinician, with reminders sent after two weeks. Recruitment and interviewing will take place until data saturation occurs (three interviews with no new shared beliefs) on the main themes. Interviews will take place at a mutually convenient time and place, ideally face to face but could be conducted over the telephone if preferred by the interviewee or if social distancing measures are still in place due to Covid-19. Further verbal and written information regarding the study will be provided prior to interview commencement and participants will be given the opportunity to ask questions. Those agreeing to take part in a face to face interview will sign a consent form in duplicate (one for the participant and one copy for the research team). Those participating in a telephone interview will be read each point of the consent form and asked to agree to each one. This will be recorded, transcribed and used as evidence of consent. Interviews will be conducted flexibly allowing for shorter interviews where necessary and participants will be reminded that the interviews can be terminated at any time. The participant can withdraw from the study at any time: data already collected with consent will be retained and used in the study. No further data will be collected, or any other research procedures carried out on or in relation to the participant. All interviews will be digitally audio recorded and transcribed verbatim by the CI or NHSG approved transcription service. The data will be stored and managed using NVivo software. Interviews will follow a semi-structured topic guide based on the COM-B behaviour change model concepts of capability, opportunity and motivation. Changes can be made to the topic guide as interviews are conducted. Data familiarisation will be by reading and rereading transcripts and by listening to the recorded interviews. Data will be analysed using iterative deductive and inductive methods combining Framework analysis and thematic analysis.

A contact will be provided for patients should they become distressed because of contact by or participation in the study. Although all data collected will stored and analysed with the strictest of confidence in line with the General Data Protection Regulations (2018), if details of any improper conduct or poor practice are disclosed the research team may be obliged to report this. The participant's GP will not be informed. Study participants will have any travel costs reimbursed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gynaecological cancer

Exclusion Criteria:

* Non-English speaking participants
* Cognitive impairment
* Terminal stage of illness
* Diagnosis through screening programmes

Ages: 18 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynaecological cancers which are female sex dependant
Study Population: Women who have been diagnosed with a gynaecological cancer
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Description of the facilitators and barriers to health seeking behaviour in women diagnosed with gynaecological cancer using semi-structured qualitative interviews. | 2 years
  Semi-structured interviews will be used to explore the facilitators and barriers to health seeking behaviour in women who have been diagnosed with a gynaecological cancer. Analysis will be narrative using both framework and thematic analysis Framework analysis will use the constructs of capability, opportunity and motivation of the COM-B behaviour tool model.

SECONDARY OUTCOMES:
Description of the perceptions of pelvic examination in women diagnosed with gynaecological cancer using semi-structured interviews. | 2 years
  Semi-structured interviews will be used to explore the perceptions to pelvic examination in women who have been diagnosed with a gynaecological cancer. Analysis will be narrative using both framework and thematic analysis Framework analysis will use the constructs of capability, opportunity and motivation of the COM-B behaviour tool model.

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Grampian, Aberdeen, Aberdeen City, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Identifiable patient data will not be shared. Interview data will be shared in a report to funders and to peer reviewed journals